CLINICAL TRIAL: NCT07091019
Title: A Real-world Chronic Myelogenous Leukemia (CML) Patient Disease Registry to Describe Patient Experience and Clinical Outcomes Among Patients With CML Receiving Approved First or Second Line Tyrosine Kinase Inhibitor (TKI) Therapy
Acronym: ASC4REAL-2
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001J1US01
Record Dates: First submitted 2025-07-14; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Chronic Myelogenous Leukemia - Chronic Phase
Keywords: CML,; CMP-CP,; ASC4REAL,; ASC4REAL-2,; chronic phase,; BCR-ABL, MMR,; TKI,; Tyrosine Kinase Inhibitor,; molecular response,; adult,; registry,; PRO,; patient reported outcome,; QOL,; quality of life,; asciminib,; bosutinib,; imatinib,; nilotinib,; dasatinib
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — asciminib; bosutinib; Dasatinib; Imatinib Mesylate; nilotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (5):
- Asciminib: Patients who started their 1L or 2L asciminib following FDA approval on or after Oct-2024 OR Patients who have exited an asciminib interventional study in US for 1L/2L CML and are continuing treatment with asciminib in routine medical care
  Interventions: Other: TKIs
- Bosutinib: Patients who started 1L or 2L bosutinib on or after Oct-2021
  Interventions: Other: TKIs
- Dasatinib: Patients who started 1L or 2L dasatinib on or after Oct-2021
  Interventions: Other: TKIs
- Imatinib: Patients who started 1L or 2L imatinib on or after Oct-2021
  Interventions: Other: TKIs
- Nilotinib: Patients who started 1L or 2L nilotinib on or after Oct-2021
  Interventions: Other: TKIs

INTERVENTIONS:
Other: TKIs — There is no treatment allocation for NIS trials. Patients administered TKI (asciminib, bosutinib, dasatinib, imatinib, nilotinib) by prescription will be enrolled.
  Other Names: Scemblix, Bosulif, Sprycel, Gleevec, Tasigna

SUMMARY:
This CML disease registry (ASC4REAL-2) aims to gather evidence on the tolerability, safety, effectiveness, and patient-reported outcomes (PRO) in real-world healthcare from patients with Ph+-CML-CP treated with TKIs approved for 1L and 2L, including prospective follow-up for 5 years identifying and describing long-term treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of Ph+-CML-CP diagnosis.
* Receiving TKI treatment (asciminib, bosutinib, dasatinib, imatinib, or nilotinib) in routine medical care either as initial therapy or after 1 prior TKI therapy.
* Receiving treatment at US and US territories (i.e., Puerto Rico) medical practice (e.g. community-based, office-based, hospital-based, academic).
* Signed informed consent form (ICF) prior to participation in the study including agreement to be tokenized so that the patient's anonymized RWD (EMRs and/or claims data) can be accessed.

Exclusion Criteria:

* Active participation in an interventional trial that may influence the management of their Ph+-CML-CP disease.
* Currently being treated with a CML TKI in 3L or beyond.
* Known presence of T315I mutation.
* Currently in TFR phase and are not on active CML TKI therapy.
* Previously received treatment with a prior stem cell transplant
* Pregnant or nursing (lactating) female.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Ph+-CML-CP who, at enrollment, are receiving 1 of 5 TKI treatments included in this registry either as initial therapy or after 1 prior TKI therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2033-05-15 (Estimated); Study Completion 2033-05-15 (Estimated)

PRIMARY OUTCOMES:
Rate of discontinuation of index TKI due to AEs | Up to 5 years
  Rate of discontinuation of index Tyrosine kinase inhibitor (TKI) due to Adverse Events (AEs)

SECONDARY OUTCOMES:
Overview of AEs | Up to 5 years
  Overview of Adverse Events (AEs) to be provided
Rate and time to switches in TKI | Up to 5 years
  Rate and time to switches in TKI to be provided
Time to discontinuation of TKI, and reasons for TKI treatment discontinuatio | Up to 5 years
  Time to discontinuation of TKI, and reasons for TKI treatment discontinuation to be provided
Distributions of Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 5 years
  PRO-CTCAE provides assessment on individual symptom/side effect related to gastrointestinal signs/symptoms (diarrhea, constipation, nausea, vomiting), cardiovascular, sleep/wake, fatigue, headache, rash, muscle spasms, myalgia, joint pain, shortness of breath/coughing/chest pain, and edema. PRO-CTC AE scores range from 0 to 4 (4 stands for very severe)
Functional Assessment of Chronic Illness Therapy - Item-GP5 (FACIT GP5) | Up to 5 years
  Functional assessment of chronic illness therapy - GP5 (FACIT-GP5): A single item question from the Functional Assessment of Cancer Therapy - General (FACT-G) that asks patients to rate the side effect bother on a 5 point Likert scale from "not at all" to "very much"
Distributions of the PRO instrument Patient-Reported Outcomes Measurement Information System Global Health-10 (PROMIS-GH-10) | Up to 5 years
  The Global Health Patient-Reported Outcomes Measurement Information System (PROMIS-10) scale is a ten-item patient-reported measure that evaluates physical, mental, and social health. From the responses to the questions, two summary scores are derived: a global physical health score and a global mental health score. These scores are then normalised to the general population using the "T-score". The T scores range from 0 to 100 points, with 0 points indicating the most severe physical and/or mental impairment and 100 points representing the best possible health status.
Distributions of the PRO instrument Medication Adherence Report Scale - 10 (MARS-10) | Up to 5 years
  Medication Adherence Report Scale - 10 (MARS-10): consists of 10 questions on forgetting, changing dosage, stopping, skipping, and taking less medication. Score ranges from 0 to 10, the higher the response the better the adherence to the medication.
Rates of molecular responses at/by specified timepoints | Up to 5 years
  Rates of molecular responses at/by specified timepoints. MR1 is defined as Breakpoint cluster region (BCR)::Abelson (ABL1) ratio ≤ 10%; MR2 as BCR::ABL1 ratio ≤ 1%; MMR as BCR::ABL1 ratio ≤ 0.1%; MR4 as BCR::ABL1 ratio ≤ 0.01%; and MR4.5 as BCR::ABL1 ratio ≤ 0.0032%.
Duration of molecular responses | Up to 5 years
  Duration of a specified molecular endpoint is defined as the time between the date of the first documented achievement of the specified molecular endpoint (on/after the first day of current TKI treatment) and the earliest date of loss of the specified molecular endpoint, treatment failure, progression to accelerated phase/blast crisis (AP/BC), or CML-related death for the patients in the analysis set who achieved molecular response at any time respectively. The duration will be censored at the last molecular assessment date while on treatment for patients who have not experienced any of the above events.
Rates of complete hematological response (CHR) at/by specified timepoints | Up to 5 years
  CHR at specified timepoints are defined as the proportion of patients who achieve response at specified timepoints. For "by" timepoints, if a patient achieves a CHR and then loses it at or before the specified timepoint, he/she will still be classified as achieving CHR by that specific timepoint.
Failure-free survival (FFS) | Up to 5 years
  FFS is defined as the time from the date of treatment start to the earliest occurrence of the following events:
  * Treatment failure as defined below based on investigator or designee assessment irrespective of entry into the TFR period
  * Confirmed loss of MMR (in 2 consecutive tests, at any time while on treatment
  * Progression to BC as defined by the WHO (Khoury et al 2022)
  * Death from any cause (including deaths observed during the survival follow-up period) For patients who have not experienced an event prior to or at the analysis cut-off date, the time will be censored at the date of last treatment or last assessment (whichever is later) or last post treatment follow-up.
Progression-free survival (PFS) | Up to 5 years
  PFS is defined as the time from the date of treatment start to the earliest occurrence of the following events:
  * progression to blastic phase
  * death from any cause
Overall survival (OS) | Up to 5 years
  Overall survival (OS) is defined as the time from the date of treatment start to the date of death from any cause or end of follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No